CLINICAL TRIAL: NCT03741062
Title: Effects of Er:YAG Photobiomodulation Therapy on Wound Healing of Human Palatal Mucosa After Connective Tissue Graft Harvesting: A Pilot Study
Brief Title: Effects of Laser Stimulation on Wound Healing of Human Palatal Tissue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Brian Wiens, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B2018:100
Record Dates: First submitted 2018-11-03; First posted 2018-11-14 (Actual); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Healing Surgical Wounds; Pain Measurement
Keywords: Laser Therapy; Low-Level Light Therapy; Periodontics; Oral Surgery; Palate; Palate, Hard

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- J. Morita AdvErl Evo Er:YAG laser (Experimental): Immediately following completion of the surgical procedure, this group will receive photobiomodulation treatment of the palatal tissue donor site with Er:YAG laser according to the parameters recommended by experts in this field and which have shown to induce maximal proliferation of human gingival fibroblasts (Energy Setting: 80 mJ, Pulse Rate: 25 Hz, Duration: 30 s).
  Interventions: Device: J. Morita AdvErl Evo Er:YAG laser
- Control (Sham Comparator): This group will receive sham treatment of the palatal tissue donor site. The laser unit will be turned off. The clinician will simulate usage of the Er:YAG laser in a manner that is indistinguishable to the patient from the experimental group.
  Interventions: Device: Control

INTERVENTIONS:
Device: J. Morita AdvErl Evo Er:YAG laser — Er:YAG laser perimeters:
  Energy = 80 mJ Pulse Rate = 25 Hz Duration = 30 s
  Arms: J. Morita AdvErl Evo Er:YAG laser
Device: Control — Sham treatment with laser unit turned off
  Arms: Control

SUMMARY:
The purpose of this study is to assess the effects of photobiomodulation (PBM) with an Er:YAG laser on the palatal donor site following subepithelial connective tissue graft (SECTG) surgery. Patient-centred outcomes and wound healing will be compared between a control group, who receives no laser treatment, and the test group receiving PBM therapy. It is hypothesized that laser stimulation will have a beneficial effect on the patient's post-operative experience as well as the healing of the tissues.

DETAILED DESCRIPTION:
The study is a randomized clinical trial comparing palatal donor sites that receive PBM with an Er:YAG laser and palatal donor sites receiving no additional treatment, following SETG surgery. A computerized randomization program will assign patients to one of two groups. Participants will be block-randomized to ensure balance between the operators.

The palate is anesthetized with 2% lidocaine (1:100000 epinephrine) by greater palatine nerve block, nasopalatine nerve block, and local infiltration. The thickness of the tissue at donor site of the palate is measured by transgingival probing ("bone sounding"). The palatal tissue is harvested from the area bordered mesially by the root of the canine and distally by the palatal root of the first molar, extending laterally to approximately 2 mm from the gingival margin and medially far enough to obtain an adequate area of tissue for the required size of the graft while ensuring not to encroach on the palatal neurovascular bundle.

A horizontal incision, corresponding to the necessary length of the graft, is made at 90 degrees to the bone approximately 2 mm from the gingival margin. Within this first incision, the scalpel is angled at approximately 135 degrees and a split-thickness dissection of the palatal tissue is extended medially. As the scalpel is advanced, the angle of the blade is further flattened until it is nearly parallel to the surface of the bone. The incision is extended until the necessary dimensions of the graft tissue are reached. Incisions are then made to the bone at the mesial, distal, and medial borders of the graft. The donor tissue is detached from the bone with a periosteal elevator and placed on a saline-soaked gauze.

The length, width, and thickness of the graft, the thickness of the remaining flap of palatal tissue, and the length of the palatal incision will be measured with digital calipers to the nearest 0.1 mm. The palatal incision will be closed with cyanoacrylate. Immediately following completion of the surgical procedure, Group A will receive PBM of the donor site and Group B will receive sham treatment with the laser unit turned off. The parameters used for PBM will be those shown to induce maximal proliferation of gingival fibroblasts using an Er:YAG laser: Energy [80 mJ], Duration [30 s], and Pulse Rate [25 Hz].

Post-operatively, both groups receive 2 g of Amoxicillin (or 600 mg of Clindamycin in cases of penicillin allergies) and the standard post-surgical instructions given to patients at the Graduate Periodontics clinic. Patients are then provided a Visual Analog Scale (VAS) questionnaire to rate their pain from 0-10 each night for 1 week and 30 Ibuprofen (200 mg) tablets.

Patients will be followed up with at 1-week, 2-week, and 6-week post-operative appointments. Photographs will be taken at all appointments. At the first appointment, participants will return their completed VAS and any remaining Ibuprofen tablets. The donor site will be examined by a clinician who did not perform the surgery and assessed according to Fickl's Modified Early-Wound Healing Index (MEHI) and Landry's Healing Index (HI). Patients will also answer a modified Oral Impacts on Daily Performance (OIDP) questionnaire. At the 2-week appointment, the palate will again be evaluated by the same operator and assessed according to the MEHI and HI. At the 6-week appointment, the donor site will be anesthetized with local infiltration of 2% lidocaine (1:100000 epinephrine), ensuring not to inject anesthetic into the tissue overlying where the graft was harvested from. Tissue thickness at the donor site will be measured via transgingival probing, in the same method as was used pre-operatively, and a histological specimen of the tissue will be harvested and placed in 10% neutral buffered formalin. Barring any ongoing post-surgical complications at this point, the patient's participation in the study is now complete.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Full Mouth Plaque Score (FMPS) < 20%
* Full Mouth Bleeding Score (FMBS) < 20%

Exclusion Criteria:

* Any contraindications for periodontal surgery,
* Anticoagulant usage
* Corticosteroid usage
* Smoking > 10 cigarettes/day.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Cholakis, FRCD(C), Study Director — University of Manitoba
Locations (1):
- Univerisity of Manitoba, College of Dentistry, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Consensus report. Mucogingival therapy. Ann Periodontol. 1996 Nov;1(1):702-6. doi: 10.1902/annals.1996.1.1.702. No abstract available. PMID 9118277
- [Background] Zucchelli G, Mounssif I. Periodontal plastic surgery. Periodontol 2000. 2015 Jun;68(1):333-68. doi: 10.1111/prd.12059. PMID 25867992
- [Background] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Background] Aguirre-Zorzano LA, Garcia-De La Fuente AM, Estefania-Fresco R, Marichalar-Mendia X. Complications of harvesting a connective tissue graft from the palate. A retrospective study and description of a new technique. J Clin Exp Dent. 2017 Dec 1;9(12):e1439-e1445. doi: 10.4317/jced.54337. eCollection 2017 Dec. PMID 29410760
- [Background] Tonetti MS, Jepsen S; Working Group 2 of the European Workshop on Periodontology. Clinical efficacy of periodontal plastic surgery procedures: consensus report of Group 2 of the 10th European Workshop on Periodontology. J Clin Periodontol. 2014 Apr;41 Suppl 15:S36-43. doi: 10.1111/jcpe.12219. PMID 24640999
- [Background] Mei CC, Lee FY, Yeh HC. Assessment of pain perception following periodontal and implant surgeries. J Clin Periodontol. 2016 Dec;43(12):1151-1159. doi: 10.1111/jcpe.12618. Epub 2016 Nov 2. PMID 27554366
- [Background] Del Pizzo M, Modica F, Bethaz N, Priotto P, Romagnoli R. The connective tissue graft: a comparative clinical evaluation of wound healing at the palatal donor site. A preliminary study. J Clin Periodontol. 2002 Sep;29(9):848-54. doi: 10.1034/j.1600-051x.2002.290910.x. PMID 12423299
- [Background] Hurzeler MB, Weng D. A single-incision technique to harvest subepithelial connective tissue grafts from the palate. Int J Periodontics Restorative Dent. 1999 Jun;19(3):279-87. PMID 10635174
- [Background] da Silva Neves FL, Silveira CA, Dias SB, Santamaria Junior M, de Marco AC, Kerbauy WD, de Melo Filho AB, Jardini MA, Santamaria MP. Comparison of two power densities on the healing of palatal wounds after connective tissue graft removal: randomized clinical trial. Lasers Med Sci. 2016 Sep;31(7):1371-8. doi: 10.1007/s10103-016-1988-6. Epub 2016 Jun 25. PMID 27344670
- [Background] Dias SB, Fonseca MV, Dos Santos NC, Mathias IF, Martinho FC, Junior MS, Jardini MA, Santamaria MP. Effect of GaAIAs low-level laser therapy on the healing of human palate mucosa after connective tissue graft harvesting: randomized clinical trial. Lasers Med Sci. 2015 Aug;30(6):1695-702. doi: 10.1007/s10103-014-1685-2. Epub 2014 Nov 6. PMID 25373688
- [Background] Pippi R. Post-Surgical Clinical Monitoring of Soft Tissue Wound Healing in Periodontal and Implant Surgery. Int J Med Sci. 2017 Jul 18;14(8):721-728. doi: 10.7150/ijms.19727. eCollection 2017. PMID 28824306
- [Background] Aoki A, Mizutani K, Schwarz F, Sculean A, Yukna RA, Takasaki AA, Romanos GE, Taniguchi Y, Sasaki KM, Zeredo JL, Koshy G, Coluzzi DJ, White JM, Abiko Y, Ishikawa I, Izumi Y. Periodontal and peri-implant wound healing following laser therapy. Periodontol 2000. 2015 Jun;68(1):217-69. doi: 10.1111/prd.12080. PMID 25867988
- [Background] Heidari M, Paknejad M, Jamali R, Nokhbatolfoghahaei H, Fekrazad R, Moslemi N. Effect of laser photobiomodulation on wound healing and postoperative pain following free gingival graft: A split-mouth triple-blind randomized controlled clinical trial. J Photochem Photobiol B. 2017 Jul;172:109-114. doi: 10.1016/j.jphotobiol.2017.05.022. Epub 2017 May 18. PMID 28549319
- [Background] Amorim JC, de Sousa GR, de Barros Silveira L, Prates RA, Pinotti M, Ribeiro MS. Clinical study of the gingiva healing after gingivectomy and low-level laser therapy. Photomed Laser Surg. 2006 Oct;24(5):588-94. doi: 10.1089/pho.2006.24.588. PMID 17069488
- [Background] Khan I, Arany P. Biophysical Approaches for Oral Wound Healing: Emphasis on Photobiomodulation. Adv Wound Care (New Rochelle). 2015 Dec 1;4(12):724-737. doi: 10.1089/wound.2014.0623. PMID 26634185
- [Background] Ozcelik O, Cenk Haytac M, Kunin A, Seydaoglu G. Improved wound healing by low-level laser irradiation after gingivectomy operations: a controlled clinical pilot study. J Clin Periodontol. 2008 Mar;35(3):250-4. doi: 10.1111/j.1600-051X.2007.01194.x. PMID 18269665
- [Background] Enwemeka CS, Parker JC, Dowdy DS, Harkness EE, Sanford LE, Woodruff LD. The efficacy of low-power lasers in tissue repair and pain control: a meta-analysis study. Photomed Laser Surg. 2004 Aug;22(4):323-9. doi: 10.1089/pho.2004.22.323. PMID 15345176
- [Background] Woodruff LD, Bounkeo JM, Brannon WM, Dawes KS, Barham CD, Waddell DL, Enwemeka CS. The efficacy of laser therapy in wound repair: a meta-analysis of the literature. Photomed Laser Surg. 2004 Jun;22(3):241-7. doi: 10.1089/1549541041438623. PMID 15315732
- [Background] de Medeiros ML, Araujo-Filho I, da Silva EM, de Sousa Queiroz WS, Soares CD, de Carvalho MG, Maciel MA. Effect of low-level laser therapy on angiogenesis and matrix metalloproteinase-2 immunoexpression in wound repair. Lasers Med Sci. 2017 Jan;32(1):35-43. doi: 10.1007/s10103-016-2080-y. Epub 2016 Sep 20. PMID 27649960
- [Background] Pourzarandian A, Watanabe H, Ruwanpura SM, Aoki A, Ishikawa I. Effect of low-level Er:YAG laser irradiation on cultured human gingival fibroblasts. J Periodontol. 2005 Feb;76(2):187-93. doi: 10.1902/jop.2005.76.2.187. PMID 15974841
- [Background] Ogita M, Tsuchida S, Aoki A, Satoh M, Kado S, Sawabe M, Nanbara H, Kobayashi H, Takeuchi Y, Mizutani K, Sasaki Y, Nomura F, Izumi Y. Increased cell proliferation and differential protein expression induced by low-level Er:YAG laser irradiation in human gingival fibroblasts: proteomic analysis. Lasers Med Sci. 2015 Sep;30(7):1855-66. doi: 10.1007/s10103-014-1691-4. Epub 2014 Nov 28. PMID 25429773
- [Background] Kong S, Aoki A, Iwasaki K, Mizutani K, Katagiri S, Suda T, Ichinose S, Ogita M, Pavlic V, Izumi Y. Biological effects of Er:YAG laser irradiation on the proliferation of primary human gingival fibroblasts. J Biophotonics. 2018 Mar;11(3). doi: 10.1002/jbio.201700157. Epub 2017 Nov 2. PMID 29045028
- [Background] Fickl S, Fischer KR, Jockel-Schneider Y, Stappert CF, Schlagenhauf U, Kebschull M. Early wound healing and patient morbidity after single-incision vs. trap-door graft harvesting from the palate--a clinical study. Clin Oral Investig. 2014 Dec;18(9):2213-9. doi: 10.1007/s00784-014-1204-7. Epub 2014 Feb 23. PMID 24562700
- [Background] Landry RG, Turnbull RS, Howley T. Effectiveness of benzydamyne HCl in the treatment of periodontal post-surgical patients. Res Clin Forums. 10:105-118, 1988.

RESULTS

PARTICIPANT FLOW:
Groups:
- J. Morita AdvErl Evo Er:YAG Laser: Immediately following completion of the surgical procedure, this group will receive photobiomodulation treatment of the palatal tissue donor site with Er:YAG laser according to the parameters recommended by experts in this field and which have shown to induce maximal proliferation of human gingival fibroblasts (Fluence: 6.3 J/cm2, Energy Setting: 80 mJ, Pulse Rate: 25 Hz, Duration: 30 s).
  J. Morita AdvErl Evo Er:YAG laser: Er:YAG laser perimeters:
  Fluence = 6.3 J/cm^2 Energy = 80 mJ Pulse Rate = 25 Hz Duration = 30 s
Period: Overall Study
Arm/Group | J. Morita AdvErl Evo Er:YAG Laser | Control
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | J. Morita AdvErl Evo Er:YAG Laser | Control | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Full Range); unit: years] | 58.5 [39 to 72] | 62.3 [38 to 74] | 60.8 [38 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Patient Discomfort as Assessed by a Visual Analogue Scale
Description: At the end of their surgical appointment, patients will be given a Visual Analogue Scale (VAS) questionnaire to rate their post-operative pain by making a mark along a 10-cm line (0 = no pain, 10 = unbearable pain) for each night of the first post-operative week. At the one-week post-operative appointment, the participants will return their VAS questionnaires and their reported post-operative discomfort for each night of the initial post-operative week will be tabulated.
Time Frame: One week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | J. Morita AdvErl Evo Er:YAG Laser | Control
Number analyzed (Participants) | 4 | 6
score on a scale
  Day 1 | 4.90 [0.2 to 9.0] | 2.45 [0.0 to 9.3]
  Day 2 | 3.30 [0.1 to 8.0] | 0.83 [0.0 to 4.3]
  Day 3 | 2.93 [0.1 to 8.0] | 0.72 [0.0 to 3.5]
  Day 4 | 2.75 [0.2 to 7.0] | 0.40 [0.0 to 1.5]
  Day 5 | 2.65 [0.2 to 7.0] | 0.32 [0.0 to 1.2]
  Day 6 | 2.65 [0.2 to 6.0] | 0.16 [0.0 to 0.5]

2. Primary Outcome: Patient Discomfort as Assessed by Analgesic Consumption
Description: At the end of their surgical appointment, patients will be provided with a bag of 30 200-mg Ibuprofen tablets. At the one-week post-operative appointment, the participants will return any remaining Ibuprofen tablets and their total analgesic consumption for the initial post-operative week will be tabulated.
Time Frame: One week
Measure: Mean (Full Range); unit: analgesic tablets
Arm/Group | J. Morita AdvErl Evo Er:YAG Laser | Control
Number analyzed (Participants) | 4 | 6
analgesic tablets | 10.5 [1.0 to 23.0] | 6.0 [0.0 to 16.0]

3. Primary Outcome: Self-Reported Patient Discomfort as Assessed by a Oral Impacts on Daily Performance Questionnaire
Description: At the one-week post-operative appointment, patients will complete a modified Oral Impacts on Daily Performance (OIDP) questionnaire to assess the effect of the palatal wound on their oral-health related quality of life during the first post-operative week. They will rate the overall frequency of disruptions that the palatal surgical site had on eating, speaking, oral hygiene, light physical work, participation in regular outings, sleeping, relaxing, smiling and laughing, their mood, and interpersonal interactions by making a mark along a 10-cm line (0 = never, 10 = constantly) for first post-operative week. When applicable, they will also rate the overall severity of the disruptions for these same categories by making a mark along a 10-cm line (0 = barely noticeable, 10 = extremely disruptive) for first post-operative week.
Time Frame: One Week
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | J. Morita AdvErl Evo Er:YAG Laser | Control
Number analyzed (Participants) | 4 | 6
score on a scale
  Frequency of Disruptions to Eating Food | 7.52 [3.0 to 9.6] | 3.65 [0.0 to 9.5]
  Severity of Disruptions to Eating Food | 5.25 [0.1 to 8.2] | 2.65 [0.1 to 5.3]
  Frequency of Disruptions to Speaking | 4.73 [0.9 to 7.3] | 1.87 [0.0 to 9.2]
  Severity of Disruptions to Speaking | 3.28 [0.1 to 7.4] | 0.55 [0.0 to 1.5]
  Frequency of Disruptions when Performing Oral Hygiene | 5.18 [1.0 to 9.1] | 4.22 [0.0 to 9.7]
  Severity of Disruptions when Performing Oral Hygiene | 4.40 [0.1 to 8.8] | 4.98 [0.2 to 9.7]
  Frequency of Disruptions when Performing Light Work | 1.30 [0.6 to 2.0] | 0.25 [0.0 to 1.0]
  Severity of Disruptions when Performing Light Work | 0.90 [0.1 to 1.9] | 0.35 [0.0 to 1.0]
  Frequency of Disruptions when Going Out | 2.95 [0.6 to 6.5] | 0.38 [0.0 to 1.7]
  Severity of Disruptions when Going Out | 2.55 [0.1 to 6.7] | 0.58 [0.1 to 1.7]
  Frequency of Disruptions While Sleeping | 6.20 [4.5 to 8.1] | 1.62 [0.0 to 5.6]
  Severity of Disruptions While Sleeping | 3.03 [0.1 to 5.3] | 2.20 [0.2 to 4.7]
  Frequency of Disruptions While Relaxing | 4.53 [2.2 to 7.0] | 0.58 [0.0 to 2.7]
  Severity of Disruptions While Relaxing | 1.33 [0.1 to 3.2] | 0.80 [0.1 to 2.5]
  Frequency of Disruptions While Smiling and Laughing | 7.77 [6.0 to 9.6] | 2.22 [0.0 to 6.8]
  Severity of Disruptions While Smiling and Laughing | 4.70 [0.1 to 7.4] | 3.20 [0.4 to 6.7]
  Frequency of Disruptions to Patient's Mood | 2.83 [0.3 to 5.0] | 2.25 [0.0 to 7.6]
  Severity of Disruptions to Patient's Mood | 1.17 [0.1 to 3.1] | 3.30 [0.3 to 7.5]
  Frequency of Disruptions to Patient's Personal Interactions | 4.23 [3.6 to 5.1] | 1.00 [0.0 to 3.9]
  Severity of Disruptions to Patient's Personal Interactions | 2.90 [0.1 to 5.1] | 1.43 [0.1 to 3.9]

4. Secondary Outcome: Healing of the Palatal Donor Site as Assessed by Histological Analysis
Description: At a six-week post-operative appointment, a histological specimen will be harvested with a tissue punch. Samples of laser-treated and non laser-treated palatal tissues will be histologically compared with respect to concentration of inflammatory cells, amount of Type I collagen present, and amount of Type III collagen present.
Time Frame: Six weeks
Reporting Status: Not Posted

5. Secondary Outcome: Healing of the Palatal Donor Site as Assessed by the Modified Early-Wound Healing Index
Description: At the one-week and two-week post-operative appointments, a clinician who did not perform the surgery and is blinded to which treatment group the patient belongs will assess the donor site according to the Modified Early-Wound Healing Index (MEHI) proposed by Fickl. The clinician will evaluate the palatal tissue donor site and rate it from 1 to 5 (1 = complete flap closure without fibrin line at the palate, 5 = incomplete flap closure with >50% necrosis of the palatal flap tissue). The progression of post-operative healing at one week and two weeks will be compared between experimental and control groups.
Time Frame: One week, Two weeks
Reporting Status: Not Posted

6. Secondary Outcome: Healing of the Palatal Donor Site as Assessed by the Healing Index
Description: At the one-week and two-week post-operative appointments, a clinician who did not perform the surgery and is blinded to which treatment group the patient belongs will assess the donor site according to the Healing Index (HI) proposed by Landry, Turnbull, and Howley. The clinician will evaluate the palatal tissue donor site and rate it from 1 to 5 (1 = very poor, 5 = excellent) based on the parameters of tissue colour, bleeding response to palpation, presence of granulation tissue, presence of suppuration, exposure of underlying connective tissue, and epithelialization along incision margins. The progression of post-operative healing at one week and two weeks will be compared between experimental and control groups.
Time Frame: One week, Two weeks
Reporting Status: Not Posted

7. Secondary Outcome: Healing of the Palatal Donor Site as Assessed by Tissue Thickness
Description: At a six-week post-operative appointment, tissue thickness at the donor site will be measured in millimetres via bone sounding with a periodontal probe. This will be compared to pre-operative measurements taken at the site.
Time Frame: Six weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the 6-week period during which the study was conducted for each patient.
Arm/Group | J. Morita AdvErl Evo Er:YAG Laser | Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 2/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | J. Morita AdvErl Evo Er:YAG Laser (N=5) | Control (N=6)
Inadequate Hemostasis at Donor Site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Proper hemostasis of the palatal site could not be achieved with cyanoacrylate alone, as specified in the study protocol. The palate had to be sutured and the patient was exited from the study, prior to collection of baseline information
Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — During the first post-operative week, a hematoma formed at the recipient site of the connective tissue graft.

LIMITATIONS AND CAVEATS:
Small sample size due to early termination of study because of COVID-19 pandemic.

Imbalanced distribution of genders between Control and Treatment groups (despite randomization).

Lack of standardization in methods for clinical measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03741062/Prot_SAP_000.pdf